CLINICAL TRIAL: NCT02089074
Title: Systematic Follow up of Drug Treatment by Pharmacists in Secondary Prevention After Transient Ischemic Attack: Adherence and Cardiovascular Events in the First Three Months
Brief Title: Systematic Follow up of Drug Treatment by Pharmacists in Secondary Prevention After Transient Ischemic Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Midt-Norge (Other); Sykehusapotekene i Midt Norge (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1224a
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Attack, Transient; Stroke
Keywords: Secondary Prevention; Pharmacists; Directive Counseling; Medication Adherence; Patient Compliance
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug use counselling (Experimental): Pharmacist conducting drug reconciliation, medication reviews and drug use counselling during hospitalisation. Follow up telephone calls 1 week, 1 month, 2 months and three months after discharge from hospital
  Interventions: Behavioral: Drug use counselling
- Control group (No Intervention): The patients in the control group receive no intervention just treatment and follow up according to national standards

INTERVENTIONS:
Behavioral: Drug use counselling
  Arms: drug use counselling

SUMMARY:
Use of drugs is an important factor in secondary prophylaxis after transient ischemic attack (TIA), but studies show that adherence to the prescribed drugs is often poor. This randomised controlled trial aims to investigate whether a systematic follow up of drug treatment using medication reconciliation, medication reviews and patient counselling by clinical pharmacists, improves adherence and/or decreases cardiovascular events the first three months and the first year after TIA. Patient satisfaction will also be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Probable or possible transient ischemic attack
* Residing in Central Norway
* Examined within 2 weeks after the onset of symptoms
* Modified Rankin Scale 3 or less and living at home
* enrolled in the MIDNOR-TIA study NCT02038725
* Informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
adherence to drug treatment in secondary prevention after TIA | 3 months
  self reporting of adherence

SECONDARY OUTCOMES:
adherence to drug treatment in secondary prevention after TIA | 1 year
  self reporting of adherence
Persistence | 3 months
  Persistence measured by control of filled prescriptions
Incidence of stroke and cardiovascular events and deaths | 3 months
  Measured by using data from national health registries
degree of disability or dependence in the daily activities | 3 months
  measured by modified Rankin Scale and indirectly by level of care
patient satisfaction | 3 months
  Measured by using data from the Norwegian Stroke Registry
Persistence | 1 year
  Persistence measured by control of filled prescriptions
Incidence of stroke and cardiovascular events and deaths | 1 year
  Measured by using data from national health registries
degree of disability or dependence in the daily activities | 1 year
  measured by modified Rankin Scale and indirectly by level of care
patient satisfaction | 1 year
  Measured by using data from the Norwegian Stroke Registry

CONTACTS AND LOCATIONS:
Overall Officials: Bent Indredavik, PhD, Prof, Study Director — Norwegian University of Science and Technology
Locations (6):
- Norway (6):
  - Ålesund Sykehus, Ålesund
  - Kristiansund Sykehus, Kristiansund
  - Levanger Sykehus, Levanger
  - Molde Sykehus, Molde
  - Namsos Sykehus, Namsos
  - St Olavs Hospital, Trondheim